CLINICAL TRIAL: NCT04335734
Title: Influence of Wrap Fixation Technique on the Results of Fundoplication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grubnik Volodymyr (Other)
Responsible Party: Sponsor-Investigator, Grubnik Volodymyr, MD, Professor, Odessa National Medical University
Organization: Odessa National Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONMedU 1
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Gastro Oesophageal Reflux Disease
Keywords: Gastro Oesophageal Reflux Disease, Nissen Fundoplication
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Fundoplication

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nissen fundoplication with fixation of the wrap (Active Comparator): In this arm, which included 87 patients we performed the following manipulations: NF was supplemented with suturing wrap to the diaphragmatic crura (52 patients) on each side using two non-absorbable stitches. In case of weak conditions of crura or short esophagus (35 patients) fundoplication wrap was sutured to the body of stomach using two non-absorbable stitches on each side. .
  Interventions: Procedure: Nissen Fundoplication with wrap fixation
- Nissen fundoplication without fixation of the wrap (Active Comparator): Arm included 51 patients, who underwent classic Nissen fundoplication without wrap fixation.
  Interventions: Procedure: Nissen Fundoplication without wrap fixation

INTERVENTIONS:
Procedure: Nissen Fundoplication with wrap fixation — Firstly, we performed left crural dissection, division of the short gastric vessels, right crural dissection, and esophageal mobilization. Then repair of HH were made by simple cruroraphy if the size of the defect was less then 10 сm² otherwise mesh for reinforcement of cruroraphy was used. Creation of the wrap was made by passing posterior fundus behind the esophagus from left to right, followed by stitching the edges of the stomach with three interrupted sutures. Wrap was fixated to both diaphragmatic crura or to the body of stomach using two non-absorbable stitches on each side.
  Arms: Nissen fundoplication with fixation of the wrap
Procedure: Nissen Fundoplication without wrap fixation — Firstly, we performed left crural dissection, division of the short gastric vessels, right crural dissection, and esophageal mobilization. Then repair of HH were made by simple cruroraphy if the size of the defect was less then 10 сm² otherwise mesh for reinforcement of cruroraphy was used. Creation of the wrap was made by passing posterior fundus behind the esophagus from left to right, followed by stitching the edges of the stomach with three interrupted sutures.
  Arms: Nissen fundoplication without fixation of the wrap

SUMMARY:
Patients who underwent anti-reflux surgery were divided into two groups. In the I group Nissen fundoplication was supplemented with suturing wrap to the crura or the body of stomach using two non-absorbable stitches on each side. Control group included patients who underwent classic Nissen fundoplication without wrap fixation. All patients were assessed before and after surgery using validated symptoms and quality of life (GERD-HRQL) questionnaires, 24-h impedance-pH monitoring and barium-swallow.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20 - 80 years;
* Gastroesophageal reflux disease as evidence by gastroscopy and pH-monitoring;
* HH type I, II

Exclusion Criteria:

* Age < 20 years and > 80 years;
* Unable to undergo laparoscopic fundoplication due to: severe comorbidities (ASA III and more), previous major surgery with severe adhesions, etc.;
* HH type III, IV;
* BMI < 16 and > 45 kg/m²;
* Pregnancy (in females);
* Oesophageal motility disorders;
* Oesophageal peptic strictures;
* Oesophageal diverticula, other types (i.e. non-reflux) of chronic esophagitis, connective tissue disorders (e.g. scleroderma);
* History of oesophageal/gastric/duodenal surgery including vagotomy;
* Relapsing course of ulcer disease/hyperacid gastritis including complicated by delayed gastric/duodenal emptying

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2012-11-01 (Actual); Primary Completion 2014-10-01 (Actual); Study Completion 2019-05-28 (Actual)

PRIMARY OUTCOMES:
Recurrence rate of hiatal hernia | 60 months
  Recurrence of hiatal hernia will be assessed by barium contrast swallow study
Slipped wrap | 60 months
  Slipped wrap will be assessed by barium contrast swallow study

SECONDARY OUTCOMES:
Quality of life and satisfaction | 60 months
  Quality of life and satisfaction will be assessed by Gastroesophageal reflux disease - health-related quality of life (GERD-HRQL) score. The scale has 11 items,each item is scored from 0 to 5. A higher score indicating a better quality of life.